CLINICAL TRIAL: NCT06421961
Title: Digital Techniques for Measuring Chronic Leg Ulcers in Peripheral Arterial Disease: Aspects of Measurement Precision and Evaluation of Wound Treatment
Brief Title: Agreement Study on AI-assisted Smartphone-based Monitoring Tool for Difficult-to-heal Ischemic Leg Ulcers
Status: Enrolling by invitation | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Louise Koch-Nielsen, Specialist nurse, PhD student, Sahlgrenska University Hospital
Other Study IDs: AW-trail20240409
Record Dates: First submitted 2024-04-15; First posted 2024-05-20 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Chronic Limb-Threatening Ischemia
Keywords: Wound Healing; Artificial Intelligence; Digital Technology
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the project is to investigate the agreement with Bland-Altman plots between an AI-supported automatic digital measurement method of wound area and depth and existing manual measurement methods in patients with arterial ulcers on the lower leg. The expectation is that the digital measurement tool can provide healthcare providers with better opportunities to objectively monitor and detect changes in the wound healing process in patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults with peripheral arterial disease.
* Arterial or arteriovenous ulcers on lower leg
* Age <18

Exclusion Criteria:

* Adults with non-ischemic ulcers,
* Purely venous ulcers,
* Purely traumatic wounds,
* Wounds resulting from non-atherosclerotic chronic vascular conditions of the lower extremity (e.g.,vasculitis, Buerger disease, radiation arteritis),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patienten seeking care and being diagnos with peripheral arterial disease and having hard to heal wounds on lower leg or foot.
Sampling Method: Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical agreement between two methods of measuring arterial wound size, we will utilize the Bland-Altman plot. | Wounds will be sequentially included until we achieve a sample size of 223 wounds within an estimated timeframe of 52 weeks.
  The size of the wound will be determined using three different measurement techniques, with images captured during a single session.
  1. Traditional Method for Area Measurement: This method utilizes a Canon EOS 700D camera and a 10 cm ruler for reference. The area is calculated using Picsara software, yielding results in square centimeters (cm²).
  2. SeeWound Method Version 1.6.4 for Area Measurement with reference card: This technique employs a specialized app to calculate the wound area in square centimeters (cm²) with the reference card.
  2. SeeWound Method Version 1.6.4 for Research: This app utilizes lidar technology to measure the area in square centimeters (cm²).
To assess the clinical agreement between two methods of measuring the depth of arterial wounds, we will utilize the Bland-Altman plot. | Wounds will be sequentially included until we achieve a sample size of 223 wounds within an estimated timeframe of 52 weeks.
  The Depth of the wound will be determined using two different measurement techniques, with measurement taken during a single session.
  1. Manual Depth Measurement with a Cotton Swab: A cotton swab is inserted into the wound to measure its depth. The measurement is taken at the deepest point and recorded in millimeters (mm).
  2. SeeWound Method Version 1.6.4 for Research: This app utilizes lidar technology to measure the depth of the wound in millimeters (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Monica Ms Pettersson, PhD, Study Director — Sahlgrenska Academy; Joakim Mr Nordanstig, PhD, Study Chair — Sahlgrenska University Hospital; Sara Ms Haile, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden